CLINICAL TRIAL: NCT02758470
Title: The Effect of Carbonic Anhydrase Inhibitors on the Pulmonary System Response to Muscle Fatigue.
Brief Title: Muscle Fatigue and Carbonic Anhydrase Inhibitors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Glen Foster, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H16-00896
Record Dates: First submitted 2016-04-20; First posted 2016-05-02 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Hypoxia
Keywords: Muscle Fatigue; Acetazolamide; Methazolamide
MeSH Terms: conditions — Hypoxia | interventions — Acetazolamide; Methazolamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acetazolamide (Experimental): Participants will be dosed 250mg acetazolamide (p.o.) three times per day for two days prior to and a single dose on the morning of the experimental day.
  Interventions: Drug: Acetazolamide
- Methazolamide (Experimental): Participants will be dosed 100mg Methazolamide (p.o.) two times per day separated by a placebo dose for two days prior to and a single dose on the morning of the experimental day. The placebo dose is used to match the timing and number of pills taken between all arms of the study.
  Interventions: Drug: Methazolamide
- Placebo (Placebo Comparator): Participants will take three placebo pills per day for two days prior to and a single dose on the morning of the experimental day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Acetazolamide — 250 mg, taken orally three times per day
  Arms: Acetazolamide
Drug: Methazolamide — 100mg, taken orally two times per day. A placebo pill will be taken between each dose of methazolamide to match the timing of doses and the number of pills between study arms.
  Arms: Methazolamide
Other: Placebo — A placebo will be taken three times per day
  Arms: Placebo

SUMMARY:
The objective of this research is to assess the effects of acetazolamide and methazolamide on respiratory and limb muscle fatigue development. A fatiguing protocol will be conducted for the respiratory and plantar flexor muscles and the difference in pressure/torque produced by supramaximal nerve stimulation used to assess muscle fatigue between conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40 years.
* Regularly physically active
* Male

Exclusion Criteria:

* current or ex-smokers
* pulmonary function <80% of predicted
* esophageal tumour or ulcer
* have had recent (<6 months) musculoskeletal injury or any surgery to the lower leg
* have contraindications to carbonic anhydrase inhibitors (eg. severe or absolute glaucoma, adrenocortical insufficiency, hepatic insufficiency, renal insufficiency, sulfa allergy or an electrolyte imbalance such as hyperchloremic acidosis)
* are obese (BMI >30 Kg/m2)
* taking diuretics, blood thinners, or anti-platelet drugs.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2016-11; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change in trans-diaphragmatic pressure generation to supramaximal phrenic nerve stimulation following inspiratory threshold loading. | Baseline, 1, 5, 10, 20, and 30 minutes following the loading protocol for each arm of the study
Change in plantar flexor muscle group torque generation to supramaximal tibial nerve stimulation following an isometric loading protocol | Baseline, 1, 5, 10, 20, and 30 minutes following the loading protocol for each arm of the study

SECONDARY OUTCOMES:
Maximal inspiratory pressure maneuvers | Baseline and immediately following loading protocol
Maximal Voluntary Contraction of the Plantar Flexor Muscle Group | Baseline and immediately following the loading protocol
Contraction time and half-relaxation time | Baseline, 1, 5, 10, 20, and 30 minutes post loading protocol

OTHER OUTCOMES:
Esophageal and Gastric Pressure | Baseline, 1, 5, 10, 20, and 30 minutes post loading protocol
Heart Rate | Baseline, 1, 5, 10, 20, and 30 minutes post loading protocol
Beat-by-beat blood pressure | Baseline, 1, 5, 10, 20, and 30 minutes post loading protocol

CONTACTS AND LOCATIONS:
Overall Officials: Glen E Foster, Ph.D., Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

REFERENCES:
- [Result] Dominelli PB, McNeil CJ, Vermeulen TD, Stuckless TJR, Brown CV, Dominelli GS, Swenson ER, Teppema LJ, Foster GE. Effect of acetazolamide and methazolamide on diaphragm and dorsiflexor fatigue: a randomized controlled trial. J Appl Physiol (1985). 2018 Sep 1;125(3):770-779. doi: 10.1152/japplphysiol.00256.2018. Epub 2018 May 24. PMID 29792554